CLINICAL TRIAL: NCT05104346
Title: Presentation and Outcomes of Acute Appendicitis During COVID Pandemic: Lessons Learned From the Middle East (Multicenter Study)
Brief Title: Presentation and Outcomes of Acute Appendicitis During COVID Pandemic
Acronym: AA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, Gastroenterology surgical center, mansoura university, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: acute appendicitis (AA)
Record Dates: First submitted 2021-10-31; First posted 2021-11-03 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Intervention Model Description: Two groups of patients were created. Patients in group I (G1) had AA prior to the era of COVID, while patients in group II (G2) had AA during COVID
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in group I (G1) had AA prior to the era of COVID (Placebo Comparator): Patients in group I (G1) had AA prior to the era of COVID
  Interventions: Procedure: appendectomy
- patients in group II (G2) had AA during COVID (Active Comparator): patients in group II (G2) had AA during COVID
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — open or laparoscopic appendectomy

SUMMARY:
Acute appendicitis (AA) is a frequent cause of acute abdominal pain in emergency rooms around the world [1]. The lifetime risk of developing AA is estimated to be about 8% [1-3]. The severe acute respiratory syndrome SARS-CoV-2 Coronavirus (COVID-19) pandemic has raised difficult situations for healthcare systems and organizations around the world, with direct and indirect implications for patient care delivery. COVID-19 causes a wide range of clinical symptoms, including fever, dry cough, myalgia, and exhaustion, with pulmonary involvement in many cases. According to the World Health Organization (WHO), The effect of the COVID-19 pandemic on acute appendicitis and surgical care is unknown due to a lack of evidence. To see how appendicitis care has changed as a result of the COVID-19 pandemic, this study compares clinical presentation, investigative modalities, treatment procedures, and outcomes before and after the pandemic.

DETAILED DESCRIPTION:
Acute appendicitis (AA) is a frequent cause of acute abdominal pain in emergency rooms around the world [1]. The lifetime risk of developing AA is estimated to be about 8% [1-3]. The SARS-CoV-2 Coronavirus (COVID-19) pandemic has raised difficult situations for healthcare systems and organizations around the world, with direct and indirect implications for patient care delivery. COVID-19 causes a wide range of clinical symptoms, including fever, dry cough, myalgia, and exhaustion, with pulmonary involvement in many cases. According to the World Health Organization (WHO), The effect of the COVID-19 pandemic on acute appendicitis and surgical care is unknown due to a lack of evidence. To see how appendicitis care has changed as a result of the COVID-19 pandemic, this study compares clinical presentation, investigative modalities, treatment procedures, and outcomes before and after the pandemic. This is a multicenter prospective cohort study that was conducted for patients presented with Acute Appendicitis (AA).

ELIGIBILITY:
Inclusion Criteria:

patients with acute appendicitis

Exclusion Criteria:

* patients with acute appendicitis less than 12 years
* malignant appendix

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1945 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
the management strategy used | one month
  the management strategy used, which included conservative or surgical management (open or laparoscopic).

SECONDARY OUTCOMES:
clinical presentation | one month
  Alverado score from 1 to 10 the worst score is 10
postoperative complications | one month
  postoperative complications have been classified by Dindo G1 TO G5
the negative appendicectomy rate. | one month
  This is normal appendix after appendectomy

CONTACTS AND LOCATIONS:
Overall Officials: Ayman El E El Nakeeb, Principal Investigator — Mansoura University, Gastrointestinal Surgery Center
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the study protocol will be available for other researcher
Supporting Information: Study Protocol
Time Frame: available for any researcher at any time
Access Criteria: elnakeebayman@yahoo.com
URL: http://www.mans.edu.eg/

REFERENCES:
- [Result] Kim CW, Lee SH. Impact of COVID-19 on the care of acute appendicitis: a single-center experience in Korea. Ann Surg Treat Res. 2021 Oct;101(4):240-246. doi: 10.4174/astr.2021.101.4.240. Epub 2021 Oct 1. PMID 34692596
- [Result] Kohler F, Muller S, Hendricks A, Kastner C, Reese L, Boerner K, Flemming S, Lock JF, Germer CT, Wiegering A. Changes in appendicitis treatment during the COVID-19 pandemic - A systematic review and meta-analysis. Int J Surg. 2021 Nov;95:106148. doi: 10.1016/j.ijsu.2021.106148. Epub 2021 Oct 23. PMID 34700020
- [Result] Zheng Z, Bi JT, Liu YQ, Cai X. The impact of COVID-19 pandemic on the treatment of acute appendicitis in China. Int J Colorectal Dis. 2022 Jan;37(1):215-219. doi: 10.1007/s00384-021-04031-4. Epub 2021 Oct 13. PMID 34647160
- [Result] Al Hashmi FY, Al Zuabi A, Hachim IY, Mannaerts GHH, Bekdache O. Conservative management of acute appendicitis in the era of COVID 19: A multicenter prospective observational study at the United Arab Emirates. Int J Surg Open. 2021 Oct;36:100389. doi: 10.1016/j.ijso.2021.100389. Epub 2021 Aug 25. PMID 34568625
- [Result] Farber ON, Gomez GI, Titan AL, Fisher AT, Puntasecca CJ, Arana VT, Kempinsky A, Wise CE, Bessoff KE, Hawn MT, Korndorffer JR Jr, Forrester JD, Esquivel MM. Impact of COVID-19 on presentation, management, and outcomes of acute care surgery for gallbladder disease and acute appendicitis. World J Gastrointest Surg. 2021 Aug 27;13(8):859-870. doi: 10.4240/wjgs.v13.i8.859. PMID 34512909
- [Result] Rudnicki Y, Soback H, Mekiten O, Lifshiz G, Avital S. The impact of COVID-19 pandemic lockdown on the incidence and outcome of complicated appendicitis. Surg Endosc. 2022 May;36(5):3460-3466. doi: 10.1007/s00464-021-08667-9. Epub 2021 Jul 26. PMID 34312724
- See also: mansoura university — http://www.mans.edu.eg/
- Available data/document: Study Protocol: COVID and acute appendicitis — http://www.mans.edu.eg/